CLINICAL TRIAL: NCT01328366
Title: A Real World Observational Study to Evaluate the Impact of Adalimumab Therapy on Quality of Life and Psychological Factors Associated With Severe Psoriasis
Brief Title: Quality of Life and Psychosocial Factors Associated With Severe Psoriasis Following Treatment With Adalimumab
Acronym: Body Image
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: pH Associates (Unknown)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-627
Record Dates: First submitted 2011-04-01; First posted 2011-04-04 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Psoriasis
Keywords: Quality of Life; Psychosocial factors
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with severe psoriasis: The participants had severe disease as defined by a total Psoriasis Area Severity Index (PASI) of 10 or more and a Dermatology Life Quality Index (DLQI) of more than 10 and had not responded to standard systemic therapies.

SUMMARY:
The impact of psoriasis on an individual's emotional and social well-being goes beyond skin symptoms of the disease. Data suggests patients with severe psoriasis experience a greater prevalence of depressive symptoms, mood disturbances, anxiety and even suicidal ideation. Given the nature of the disease and the treatment failures which are required before a patient commences a biologic therapy such as adalimumab, the patient's mental health at initiation of biologics is an important consideration for clinicians. This study seeks to explore if adalimumab treatment of psoriasis leads to a positive impact on psychosocial factors and disease-related quality of life.

DETAILED DESCRIPTION:
This was a multi-center, prospective, post-marketing observational study of participants with severe chronic plaque psoriasis who began adalimumab therapy in the United Kingdom. Although 153 participants enrolled in the study, data was only analyzed on 143 individuals and there were no interventions or changes to participant management for the study. Prior to initiating adalimumab therapy (baseline), the Dermatology Life Quality Index (DLQI), Self-Administered Psoriasis Area Severity Index (SAPASI), Hospital Anxiety and Depression Scale (HADS), Cutaneous Body Image (CBI) scale, Short Form 12 (SF-12) Health Survey, Female Sexual Function Index (FSFI) (female participants) and International Index of Erectile Function (IIEF) (male participants) questionnaires were completed by participants and at 4 weeks, 16 weeks and 6 months following initiation.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible for adalimumab as determined by the National Institute for Health and Clinical Excellence (NICE) criteria
* Participants had severe psoriasis as defined by a Psoriasis Area Severity Index (PASI) of 10 or more and a Dermatology Life Quality Index (DLQI) of more than 10
* Participant's psoriasis did not respond to standard systemic therapies, to include: ciclosporin, methotrexate, and psoralen and long-wave ultraviolet radiation; or the participant was intolerant of or had a contraindication to these treatments

Exclusion Criteria:

* Participants were previously treated with another biologic therapy
* Participants were unable or unwilling to complete the study questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary Care Outpatients
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Pumford, MD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Severe Psoriasis
Started | 153
Completed | 143
Not Completed | 10
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Population: The participants had severe disease as defined by a total Psoriasis Area Severity Index (PASI) of 10 or more and a Dermatology Life Quality Index (DLQI) of more than 10 and had not responded to standard systemic therapies. Baseline demographic data was not available for all participants.
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.0 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 87

OUTCOME MEASURES:

1. Primary Outcome: Dermatology Life Quality Index (DLQI) Scores
Description: The Dermatology Life Quality Index (DLQI) was a participant-reported questionnaire used to measure the health-related quality of life (QOL) of adults suffering from a skin disease. Scores ranged from 0-30, a higher score indicating a greater impact on a participant's QOL. Data are reported as the mean DLQI score ± standard deviation.
Time Frame: Baseline; 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Participants who completed the DLQI questionnaire at Baseline, 4 Week, 16 Week, or their 6 Month assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 134
units on a scale
  Baseline | 17.25 (6.51)
  4 Weeks (n=43) | 8.65 (6.51)
  16 Weeks (n=80) | 4.51 (5.88)
  6 Months (n=100) | 3.65 (6.41)

2. Primary Outcome: Mean Change in Dermatology Life Quality Index (DLQI) Scores From Baseline
Description: The Dermatology Life Quality Index (DLQI) was a participant-reported questionnaire used to measure the health-related quality of life (QOL) of adults suffering from a skin disease. Scores ranged from 0-30, a higher score indicated a greater impact on a participant's QOL. "Responders" to adalimumab had a ≥5 point reduction in DLQI scores or DLQI score of 0. Data are reported as the mean DLQI score ± standard deviation.
Time Frame: 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Participants who completed the DLQI questionnaire at baseline and at the 4 Week, 16 Week, or 6 Month assessment. Participants who did not complete a Baseline and 4 Week, 16 Week, or 6 Month assessment were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 134
units on a scale
  4 Weeks (n=38) | -9.95 [-12.07 to -7.82]
  16 Weeks (n=76) | -13.03 [-14.69 to -11.36]
  6 Months (n=94) | -13.63 [-15.29 to -11.97]

3. Secondary Outcome: Self-assessed Psoriasis Area and Severity Index (SAPASI) Scores
Description: The Self-assessed Psoriasis Area and Severity Index (SAPASI) questionnaire was used to objectively measure the severity of a participant's psoriasis, taking into account the area of psoriasis legions on the body and the characteristics of these legions (redness, thickness, scaliness). Scores ranged from 0-72, a higher score indicated more severe psoriasis. Data are reported as the mean SAPASI score ± standard deviation.
Time Frame: Baseline; 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Participants who completed the SAPASI questionnaire at Baseline, 4 Weeks, 16 Weeks, or their 6 Month assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 128
units on a scale
  Baseline (n=128) | 21.02 (11.42)
  4 Weeks (n=43) | 7.37 (7.13)
  16 Weeks (n=78) | 4.42 (6.54)
  6 Months (n=97) | 4.41 (7.81)

4. Secondary Outcome: Mean Change in Self-assessed Psoriasis Area and Severity Index (SAPASI) Scores From Baseline
Description: The Self-assessed Psoriasis Area and Severity Index (SAPASI) questionnaire was used to objectively measure the severity of a participant's psoriasis, taking into account the area of psoriasis legions on the body and the characteristics of these legions (redness, thickness, scaliness). Scores ranged from 0-72, a higher score indicated more severe psoriasis. Data are reported as the mean change in SAPASI score ± standard deviation.
Time Frame: 4 weeks, 16 weeks, and 6 months after adalimumab initiation
Population: Participants who completed the SAPASI questionnaire at Baseline, 4 Weeks, 16 Weeks, or their 6 Month assessment. Participants who did not complete a Baseline and 4 Week, 16 Week, or 6 Month assessment were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 128
units on a scale
  4 Weeks (n=35) | -16.41 [-20.18 to -12.65]
  16 Weeks (n=72) | -18.79 [-21.78 to -15.80]
  6 Months (n=87) | -17.34 [-19.94 to -14.74]

5. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Scores
Description: The Psoriasis Area and Severity Index (PASI) questionnaire was used by the clinical staff to measure the severity of a participant's psoriasis, taking into account the area of psoriasis legions on the body and the characteristics of these legions (redness, thickness, scaliness). Scores ranged from 0-72, a higher score indicated more severe psoriasis. Data are reported as the mean PASI score ± standard deviation.
Time Frame: Baseline; 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Participants who completed the PASI questionnaire at Baseline, 4 Weeks, 16 Weeks, or their 6 Month assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 124
units on a scale
  Baseline | 16.98 (8.47)
  4 Weeks (n=24) | 5.52 (4.48)
  16 Weeks (n=81) | 3.42 (5.31)
  6 Months (n=91) | 2.38 (3.98)

6. Secondary Outcome: Mean Change in Psoriasis Area and Severity Index (PASI) Scores From Baseline
Description: The Psoriasis Area and Severity Index (PASI) questionnaire was used by the clinical staff to measure the severity of a participant's psoriasis, taking into account the area of psoriasis legions on the body and the characteristics of these legions (redness, thickness, scaliness). Scores range from 0-72, a higher score indicating more severe psoriasis. Data are reported as the mean change in PASI score ± standard deviation.
Time Frame: 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Participants who completed the PASI questionnaire at Baseline, 4 Weeks, 16 Weeks, or their 6 Month assessment. Participants who did not complete a Baseline and 4 Week, 16 Week, or 6 Month assessment were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 124
units on a scale
  4 Weeks (n=24) | -10.90 [-14.05 to -7.75]
  16 Weeks (n=80) | -13.93 [-15.90 to -11.96]
  6 Months (n=89) | -13.99 [-15.75 to -12.22]

7. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) Scores
Description: The Hospital Anxiety and Depression Scale (HADS) was a patient-reported questionnaire used to assess the level of anxiety and depression in the setting of a hospital medical outpatient clinic. The anxiety and depression subscales each have a range from 0-21, higher scores indicated higher levels of anxiety and depression, respectively. Data are reported as the mean anxiety or depression score ± standard deviation.
Time Frame: Baseline; 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Participants who completed the HADS questionnaire at Baseline, 4 Week, 16 Week, or their 6 Month assessment. HADS-A refers to the anxiety, while HADS-D refers to the depression portion of the survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 132
units on a scale
  HADS-A Baseline | 9.63 (4.70)
  HADS-A 4 Weeks (n=43) | 8.21 (4.95)
  HADS-A 16 Weeks (n=80) | 6.65 (4.22)
  HADS-A 6 Months (n=100) | 6.00 (4.29)
  HADS-D Baseline | 7.08 (4.46)
  HADS-D 4 Weeks (n=43) | 6.19 (4.68)
  HADS-D 16 Weeks (n=80) | 4.18 (3.67)
  HADS-D 6 Months (n=100) | 3.43 (3.63)

8. Secondary Outcome: Mean Change in Hospital Anxiety and Depression Scale (HADS) Scores From Baseline
Description: The Hospital Anxiety and Depression Scale (HADS) was a patient-reported questionnaire used to assess the level of anxiety and depression in the setting of a hospital medical outpatient clinic. The anxiety and depression subscales each have a range from 0-21, higher scores indicated higher levels of anxiety and depression, respectively. Data are reported as the mean change in anxiety or depression score ± standard deviation.
Time Frame: 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Participants who completed the HADS questionnaire at baseline and at the 4 Week, 16 Week, or 6 Month assessment. Participants who did not complete a Baseline and 4 Week, 16 Week, or 6 Month assessment were not included in the analysis. HADS-A refers to the anxiety, while HADS-D refers to the depression portion of the survey.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 132
units on a scale
  HADS-A 4 Weeks (n=36) | -1.56 [-2.87 to -0.24]
  HADS-A 16 Weeks (n=74) | -2.81 [-3.70 to -1.92]
  HADS-A 6 Months (n=93) | -3.32 [-4.17 to -2.48]
  HADS-D 4 Weeks (n=36) | -1.58 [-2.83 to -0.34]
  HADS-D 16 Weeks (n=74) | -2.68 [-3.56 to -1.79]
  HADS-D 6 Months (n=93) | -3.14 [-3.97 to -2.31]

9. Secondary Outcome: Cutaneous Body Image Scale (CBI) Scores
Description: The Cutaneous Body Image (CBI) Scale was a participant-reported questionnaire used to measure a participant's satisfaction with their hair, nails, and skin. Scores range from 0-9, higher scores indicated a higher level of satisfaction. Data are reported as the mean CBI score ± standard deviation.
Time Frame: Baseline; 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Participants who completed the CBI questionnaire at Baseline, 4 Week, 16 Week, or their 6 Month assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 134
units on a scale
  Baseline | 2.73 (1.83)
  4 Weeks (n=42) | 4.38 (1.92)
  16 Weeks (n=80) | 5.58 (1.85)
  6 Months (n=100) | 6.16 (1.98)

10. Secondary Outcome: Mean Change in Cutaneous Body Image (CBI) Scale Scores From Baseline
Description: The Cutaneous Body Image (CBI) Scale was a participant-reported questionnaire used to measure a participant's satisfaction with their hair, nails, and skin. Scores range from 0-9, higher scores indicated a higher level of satisfaction. Data are reported as the mean change in CBI score ± standard deviation.
Time Frame: 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Participants who completed the CBI questionnaire at baseline and at the 4 Week, 16 Week, or 6 Month assessment. Participants who did not complete a Baseline and 4 Week, 16 Week, or 6 Month assessment were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 134
units on a scale
  4 Weeks (n=37) | 2.05 [1.28 to 2.82]
  16 Weeks (n=76) | 2.83 [2.29 to 3.38]
  6 Months (n=95) | 3.45 [2.92 to 3.97]

11. Secondary Outcome: 12-item Short Form Survey (SF-12) Score
Description: The 12-item Short Form Survey (SF-12) was a participant-reported questionnaire use to measure the functional health and well-being of a participant to include both physical and mental health domains. Scores range from 0-100 for each domain, higher scores indicated better physical or mental health. Data are reported as the mean SF-12 score physical or mental ± standard deviation.
Time Frame: Baseline; 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Participants who completed the SF-12 questionnaire at Baseline, 4 Week, 16 Week, or their 6 Month assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 127
units on a scale
  SF-12 Physical Baseline | 43.08 (11.61)
  SF-12 Physical 4 Weeks (n=42) | 46.38 (11.35)
  SF-12 Physical 16 Weeks (n=74) | 50.53 (8.50)
  SF-12 Physical 6 Months (n=97) | 49.53 (10.05)
  SF-12 Mental Baseline | 41.23 (11.25)
  SF-12 Mental 4 Weeks (n=42) | 45.50 (10.53)
  SF-12 Mental 16 Weeks (n=74) | 46.84 (11.12)
  SF-12 6 Months (n=97) | 49.22 (10.15)

12. Secondary Outcome: Change in 12-item Short Form Survey (SF-12) Score From Baseline
Description: The 12-item Short Form Survey (SF-12) was a participant-reported questionnaire use to measure the functional health and well-being of a participant to include both physical and mental health domains. Scores range from 0-100 for each domain, higher scores indicated better physical or mental health. Data are reported as the mean change SF-12 score physical or mental ± standard deviation.
Time Frame: 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Participants who completed the SF-12 questionnaire at baseline and at the 4 Week, 16 Week, or 6 Month assessment. Participants who did not complete a Baseline and 4 Week, 16 Week, or 6 Month assessment were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 127
units on a scale
  SF-12 Physical 4 Weeks (n=36) | 4.60 [1.77 to 7.44]
  SF-12 Physical 16 Weeks (n=69) | 6.84 [4.60 to 9.08]
  SF-12 Physical 6 Months (n=89) | 6.46 [4.39 to 8.54]
  SF-12 Mental 4 Weeks (n=36) | 4.96 [1.21 to 8.71]
  SF-12 Mental 16 Weeks (n=69) | 6.10 [3.32 to 8.88]
  SF-12 Mental 6 Months (n=89) | 6.47 [4.11 to 8.84]

13. Secondary Outcome: Female Sexual Function Index (FSFI) Score
Description: The Female Sexual Function Index (FSFI) was a participant-reported questionnaire used to measure a female's sexual function. Scores range from 2-36, higher scores indicated better sexual function. Data are reported as the mean FSFI score ± standard deviation.
Time Frame: Baseline; 16 weeks, and 6 months following adalimumab initiation
Population: Female participants who completed the FSFI questionnaire at Baseline, 4 Week, 16 Week, or their 6 Month assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 36
units on a scale
  Baseline | 15.77 (10.50)
  16 Weeks (n=18) | 18.65 (12.70)
  6 Months (n=26) | 20.73 (11.70)

14. Secondary Outcome: Mean Change in Female Sexual Function Index (FSFI) Score From Baseline
Description: The Female Sexual Function Index was a participant-reported questionnaire used to measure a female's sexual function. Scores range from 2-36, higher scores indicated better sexual function. Data are reported as the mean change in FSFI score ± standard deviation.
Time Frame: 4 week, 16 weeks, and 6 months following adalimumab initiation
Population: Female participants who completed the FSFI questionnaire at baseline and at the 4 Week, 16 Week, or 6 Month assessment. Participants who did not complete a Baseline and 4 Week, 16 Week, or 6 Month assessment were not included in the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 36
units on a scale
  4 Weeks (n=4) | 3.78 [-8.76 to 16.31]
  16 Weeks (n=15) | 0.53 [-5.73 to 6.80]
  6 Months (n=21) | 4.72 [1.33 to 8.11]

15. Secondary Outcome: International Index of Erectile Function Score
Description: The International Index of Erectile Function (IIEF) was a participant-reported questionnaire used to measure a male's erection function. Scores range from 5-75, higher scores indicated better erection quality. Data are reported as the mean IIEF score ± standard deviation.
Time Frame: Baseline; 4 weeks, 16 weeks, and 6 months following adalimumab initiation
Population: Male participants who completed the IIEF questionnaire at Baseline, 4 Week, 16 Week, or their 6 Month assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Severe Psoriasis
Number analyzed (Participants) | 64
units on a scale
  Baseline | 56.05 (19.20)
  4 Weeks (n=24) | 58.33 (13.80)
  16 Weeks (n=36) | 60.61 (17.50)
  6 Months (n=47) | 54.43 (22.90)

ADVERSE EVENTS:
Time Frame: From informed consent to completion of final study questionnaire
Arm/Group | Participants With Severe Psoriasis
Serious Adverse Events (participants affected / at risk) | 0/143
Other Adverse Events (participants affected / at risk) | 5/143
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Severe Psoriasis (N=143)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Headache (Nervous system disorders) | 1
Rash pustular (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.